CLINICAL TRIAL: NCT05275829
Title: Traditional Face-to-Face Versus Distance Learning of Basic Suturing Skills in Novice Learners
Brief Title: Face-to-Face Versus Distance Learning of Basic Suturing Skills
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Ahmad Zaghal, Assistant Professor of Clinical Speciality, American University of Beirut Medical Center
Other Study IDs: SBS-2020-0378
Record Dates: First submitted 2022-02-24; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Educational Problems
Keywords: Medical Education; Suturing Skills; Face-to-Face learning; Distance Learning; Pandemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Face-to-Face learning of simple interrupted suturing: * The students watched a video demonstrating simple interrupted suturing, with the instructor commenting on the steps.
  * The students then watched the video again.
  * The instructor then demonstrated the procedure for the students.
  * The students then practiced suturing with immediate and specific feedback provided by the instructor until he and the students were satisfied with the performance.
- Study group: Distance learning (tele simulation) of simple interrupted suturing: * The instructor ran the interactive tele simulation sessions utilising web-based video-conferencing technology (WebEx platform). The students used their personal smartphones or laptops with audio-video capabilities. The instructor ran the session through his smartphone.
  * The instructor shared a video demonstrating simple interrupted suturing while commenting on the steps (the same video used in the control group).
  * The instructor then ran the video again for the students.
  * The instructor then demonstrated the skill for the students by turning on his camera.
  * The students then practiced suturing, and periodically turned on their cameras to receive live and specific feedback from the instructor on their performance, until the instructor and the students were satisfied.
  * No face-to-face interactions between the students and the instructor.
  Interventions: Other: Tele simulation

INTERVENTIONS:
Other: Tele simulation — Interactive tele simulation sessions utilising web-based video-conferencing technology (WebEx platform).
  Groups: Study group: Distance learning (tele simulation) of simple interrupted suturing

SUMMARY:
The main objective of this study is to determine the acceptability and effectiveness of Distance Learning (DL) of basic suturing skills in novice learners.

A prospective randomized controlled trial involving 118 pre-medical and medical students with no previous experience in suturing was conducted. Participants were randomized into two groups for learning simple interrupted suturing: F-F and DL groups (59 students in each group) . Evaluation was conducted by two independent assessors. Agreement between the assessors was calculated, and performance scores of the participants were compared between the two groups.

All the participants demonstrated their ability to place three interrupted sutures, with no significant difference in the performance between the two groups. All the respondents positively rated the teaching sessions, found them useful and enjoyable.

Distance learning of basic suturing is as effective as the face-to-face approach in novice learners

DETAILED DESCRIPTION:
At our hospital, during the initial lock-down period in March and April 2020, all medical students' clinical clerkships were temporarily cancelled, and their educational activities switched to web-based remote learning, utilizing teleconferencing and commercially available web-based interactive clinical modules. Teaching surgical technical skills, such as basic suturing, presented itself as a more challenging component of the clinical education under these unusual circumstances as compared to teaching cognitive skills and knowledge, which raised questions and concerns around the effectiveness and acceptability of distance learning of basic surgical skills.

In this study, the investigators aimed to compare the effectiveness and retention of distance learning to the traditional face-to-face learning of basic (simple interrupted) suturing in novice learners. This study entails a prospective randomized trial involving two arms (traditional face-to-face versus distance learning of basic simple interrupted suturing) in pre-medical students as well as first and second year medical students at the American University of Beirut (AUB). Immediately after the teaching session as part of research, two independent surgeons assessed the students' simple interrupted suturing performance using a validated checklist and OSATS global rating.

The difference in performance was used to determine the effectiveness of distance learning of basic suturing as compared to the traditional instructional method. In addition, the students in both groups were asked to complete a questionnaire (immediately after the teaching session) to investigate their satisfaction and confidence.

ELIGIBILITY:
Inclusion Criteria:

* Pre-medical, first, and second-year medical students with no previous experience in suturing.

Exclusion Criteria:

* Previous experience in suturing.Refusal of enrolment.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pre-medical, first, and second-year medical students from a four-year Doctor of Medicine graduate-entry programme. Premedical students include senior biology, medical laboratory, and nutrition students. All participants had no previous experience with suturing. Basic suturing is one of the educational activities of the third-year medical students, before which students are not normally exposed to basic suturing skills teaching sessions. The participants were recruited via an email sent to all the potential candidates for participation in this study.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Assessment of suturing skills in medical students via checklist | immediately after the intervention(suturing session)
  The adopted ten-item checklist for assessing suturing skills in medical studentS differentiated between novice and expert performances and showed a narrow variation in the scores provided by three independent expert assessors.
  Overall performance scores were calculated based on the formula used by the same authors: "cutoff time (seconds) - completion time (seconds) - (10 x sum of errors)" with higher scores indicating better performance

SECONDARY OUTCOMES:
Assessment of suturing skills in medical students via OSATS | immediately after the intervention(suturing session)
  OSATS is a validated observational assessment tool also used in medical students. It comprises of seven performance domains whereby learners are scored on a 5-point Likert scale on proper tissue handling, efficiency and economy of movements, instrument handling, suture handling, flow of the procedure, knowledge of the steps of the procedure, overall appearance of the suture, in addition to an overall assessment of the performance; higher scores indicate better performance

OTHER OUTCOMES:
Questionnaire that assesses confidence and satisfaction | immediately after the intervention( suturing session)
  The students were asked, on voluntary basis, to electronically fill a brief anonymous questionnaire after the completion of their respective sessions to evaluate their satisfaction (acceptability), confidence levels, and attitudes towards the instructional method they experienced (Figure 4). We followed the AMEE's guide No.87 (Artino et-al, 2014) recommendations for the survey items development, making sure to use clear self-explanatory language, avoid using negative-worded sentences, and include verbal labels for all the Likert-scale responses of the closed-ended items. We have also included three open-ended questions to gain a more detailed grasp of the students' perceptions of their learning experience.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Zaghal, MD, MSc, FACS, FEBPS, Principal Investigator — American University of Beirut Medical Center ; Department of Surgery
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are not publicly available due to the Institutional Review Board requirements but are available from the corresponding author upon a reasonable request.